CLINICAL TRIAL: NCT01487447
Title: Customized Acoustic Stimulation for the Treatment of Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSMT003 HS# 2006-5187
Record Dates: First submitted 2011-12-02; First posted 2011-12-07 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2018-07

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: Customized sound
- Control (Active Comparator)
  Interventions: Other: Regular Masker

INTERVENTIONS:
Other: Customized sound — treatment with customized sound therapy
  Arms: Intervention
Other: Regular Masker — treatment with white noise
  Arms: Control

SUMMARY:
The purpose of this study is to determine the efficacy of a customized sound therapy in reducing tinnitus loudness and increasing the residual inhibition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male or female
* Tinnitus present for 6 months or more
* Adequate command of English

Exclusion Criteria:

* Active illicit drug use, alcohol dependence
* Treatable cause of tinnitus
* History of psychosis
* Subjects on medications known to cause tinnitus (aspirin, ibuprofen, naproxen) which could not be stopped will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in score of tinnitus loudness | 0, 1 minute; 1 hour; 1, 2, 4 and 6 months
Change in score of tinnitus annoyance | 0, 1 minute; 1 hour; 1, 2, 4 and 6 months
Change in residual inhibition | 1 minute; 1 hour; 1, 2, 4 and 6 months
Change in score of Tinnitus Handicap Inventory (THI) | 0, 1, 2, 4 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine Medical Center, Orange, California, United States